CLINICAL TRIAL: NCT00527969
Title: Cognitive, Emotional, Physical, and Psychosocial Effects of Three Weeks' Prospective Double-Blind Placebo Controlled Cross-Over Exposure to Panax Quinquefolius L (REMEMBER-fX), With Optional Six Months' Open Label Follow-up
Brief Title: Cognitive, Emotional, Physical and Psychosocial Effects of Panax Quinquefolius L
Acronym: REMEMBER-fX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CV Technologies (Industry)
Organization: Afexa Life Sciences Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HT1001-2006-2
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Memory; Learning; Attention; Cognition; Well-Being
Keywords: American ginseng extract; Panax quinquefolius; Memory enhancement; Cognitive function; Working memory; Declarative memory; Psychomotor speed; Executive skills; Psychosocial adaptation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: HT1001 extract of Panax quinquefolius L

SUMMARY:
The purpose of this study is to determine the efficacy and safety of REMEMBER-fX (HT1001, an extract of Panax quinquefolius) in a human sample using standard clinical neuropsychological instruments and side effects rating scales.

DETAILED DESCRIPTION:
Panax ginseng has been used in Asia for thousands of years to improve vitality, wakefulness, respiration, angina, nausea, attention, memory, and diminished libido. More recently, Panax extracts have become one of the most popular commercial herbal dietary supplements in the West as well. Unfortunately, a limited understanding of the bioactive ingredients within the Panax extracts resulted in a wide spectrum of available products with no guidelines for standardization. The lack of standardization undermined any legitimate attempt to validate the claimed health benefits of the extracts. However, recent advances in the identification, quantification, and standardization of extract components with demonstrated systemic and neurological actions in animals have created a novel opportunity for the controlled clinical investigation of some Panax extracts.

A significant improvement in the standardization of Panax extracts occurred approximately 20 years ago with the introduction of a 4% minimum ginsenoside content in a formulation of Panax ginseng C V Meyer under the trademark G115 by Pharmaton in Lugano Switzerland. This prompted a series of investigations of short-term cognitive, physical, emotional, and psychosocial benefits from a single dose of G115. Idiosyncratic cognitive gains were reported, but no reliable benefits were observed in physical, emotional, or psychosocial status. Several studies have examined the cognitive, physical, emotional, and psychosocial benefits from sustained exposure to G115, but these studies are few in number and often failed to include standardized behavioural measures or controlled Panax extracts.

Over the past five years, refinements in high pressure liquid chromatography (HPLC) have allowed greater precision in Panax constituent analysis, with significant implications to the investigation of the safety and efficacy of Panax extracts in human populations. HPLC has been used to identify and quantify several promising neuroactive ginsenosides that are likely relevant to the human bioactive effect of Panax extracts. Most notable are the Rg1 and Rb1 ginsenosides from Panax quinquefolius L which show a number of interesting in vitro effects on animal tissue from the central nervous system that have led to several positive results from studies of animal learning. Most significant, however, was the introduction of HT1001, a precisely standardized proprietary combination of Rg1 and Rb1 ginsenosides developed by CV Technologies in Edmonton, Alberta, Canada. Each product lot of HT1001 from CV Technologies is tested to ensure consistency of the ginsenoside composition. The introduction of a commercial product with a precise standardized composition of Rb1 and Rg1 has created a unique opportunity for investigating the safety and efficacy of Panax extracts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between the age of 35 - 75
* Women of child bearing capacity who agree to use an acceptable form of birth control during the trial (i.e. oral contraception, reliable use of a double-barrier method (e.g. condom and diaphragm, condom and foam, condom and sponge), IUD or tubal ligation)
* Achievement Test (WRAT-III) score greater than 70 with a reading level within normal limits as defined by a Wide Range
* Willing to adhere to the requirements of the protocol, including availability for follow-up visits
* Willing and able to sign written informed consent

Exclusion Criteria:

* Medical conditions;
* HIV/AIDS
* Malignancy (under active observation or treatment)
* Unstable cardiovascular disease (physician visit or hospitalization for unstable cardiovascular disease in the last 6 mo.)
* Renal Abnormalities (serum creatinine known to be > 200umol/L)
* Acute or active chronic liver disease
* Diabetes
* Neurologic or psychiatric disease (progressive or currently under treatment)
* Active tuberculosis
* Multiple sclerosis
* Bleeding disorders

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2007-07

PRIMARY OUTCOMES:
Use of HT1001 will improve objective measures of psychomotor speed, sustained attention, working memory, declarative memory, and or executive skills. | 3 weeks

SECONDARY OUTCOMES:
Use of HT1001 will be associated with no cognitive or physical adverse effects. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scot E Purdon, PhD, Principal Investigator — Department of Psychiatry, University of Alberta
Locations (1):
- PNL, Edmonton, Alberta, Canada